CLINICAL TRIAL: NCT04844333
Title: Effect of Extubation Under Deep Anesthesia on Emergence Agitation of Nasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, Chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH9H-2020-T414-2
Record Dates: First submitted 2021-04-05; First posted 2021-04-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extubation under deep anesthesia (Experimental): When the patient is in sedation or anesthesia state, including no body movement, bispectral index 60-70, spontaneous breathing recovery, VT ≥ 5ml / kg, respiratory rate 10-20 times / min, regular rhythm, PetCO2 < 45mmhg, regular waveform, stable circulation, the endotracheal tube is removed.
  Interventions: Other: Extubation under deep anesthesia
- Awake extubation (No Intervention): When the patient is in awake state, including bispectral index >70, spontaneous breathing recovery, VT ≥ 5ml / kg, respiratory rate 10-20 times / min, regular rhythm, PetCO2 < 45mmhg, regular waveform, the cough and swallowing reflex are obvious and the circulation is stable, the endotracheal tube is removed.

INTERVENTIONS:
Other: Extubation under deep anesthesia — When the patient in sedation or anesthesia state, no body movement, bispectral index 60-70, spontaneous breathing recovery, VT ≥ 5ml / kg, respiratory rate 10-20 times / min, regular rhythm, PetCO2 < 45mmhg, regular waveform, stable circulation, the patient is in deep anesthesia state, and the endotracheal tube is removed.
  Arms: Extubation under deep anesthesia

SUMMARY:
This study analyzed the relationship between extubation timing and Emergence agitation in 18-60 years old adults undergoing nasal surgery, such as nasal septum correction, endoscopic sinus surgery, and nasal bone fracture reduction. The number of agitation, sedation score, pain score, operation method, analgesic drugs and other data were recorded to analyze the effect of deep anesthesia extubation on agitation in patients with nasal surgery. It also provides a clinical basis for the prevention and treatment of agitation during the recovery period of such operations in adults.

DETAILED DESCRIPTION:
Nasal surgery is an operation with a high proportion of pain and agitation found in the clinical medical treatment of our hospital. Although the operation time is short, the operation trauma is small, and it does not involve important organs and blood vessels, the clinical observation shows that the incidence of agitation in such patients after operation is high, and the degree of pain varies greatly. Many studies have analyzed the related risk factors of agitation in the wake-up period of adult nasal surgery, and believe that the existence of postoperative endotracheal tube is the main risk factor. However, there is a lack of prospective randomized controlled study on the timing of postoperative extubation in patients with nasal surgery. Therefore, this study analyzes the impact of extubation timing on postoperative agitation, so as to clarify the correlation between postoperative agitation and extubation timing and possible protective factors, which is helpful to early prediction, prevention and treatment, and reduce the incidence of postoperative EA in patients with nasal surgery.

ELIGIBILITY:
Inclusion Criteria:

ASA grade I-II Age 18-60 Patients undergoing selective general anesthesia for the correction of septum, endoscopic sinus surgery, bone fracture reconstruction, resection of sinus tumor, augmentation of nose and other nasal surgery Subjects voluntarily participate in the study and sign informed consent

Exclusion Criteria:

History of mental and neurological diseases; History of chronic pain or long-term use of opioids and other analgesics; History of respiratory diseases, severe pulmonary dysfunction and airway hyperresponsiveness; History of severe hypertension and cardiovascular disease; Pregnant women; Patients with severe primary diseases such as liver, kidney and hematopoietic system; patients with abnormal liver function (ALT, AST and TBIL exceeding 1.5 times the upper limit of normal value) or renal dysfunction (creatinine and urea nitrogen exceeding 1.5 times the upper limit of normal value) History of alcohol or drug abuse; History of epilepsy or a recent epilepsy; Obese patients, BMI ≥ 30kg / m2, or with sleep apnea; In addition to the above, the researchers judged that they were not suitable to participate in this clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
The incidence of Emergence Agitation during recovery | During recovery period after Nasal Surgery，an average of one and a half hours
  The incidence of Emergence Agitation during recovery

CONTACTS AND LOCATIONS:
Overall Officials: jingjie Li, Ph.D, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (3):
- China (3):
  - Shanghai9 Hospital, Shanghai, Shanghai Municipality
  - Shanghai ninth people's hospital, Shanghai
  - Shanghai No.9 People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suo L, Lu L, Li J, Qiu L, Liu J, Shi J, Sun Z, Lao W, Zhou X. The effect of deep and awake extubation on emergence agitation after nasal surgery: a randomized controlled trial. BMC Anesthesiol. 2024 May 18;24(1):177. doi: 10.1186/s12871-024-02565-y. PMID 38762729